CLINICAL TRIAL: NCT06801925
Title: Evaluating the Effectiveness and Acceptability of a GPT-4o and RAG-Based Voice Chatbot for Depression Screening Using PHQ-9
Acronym: GPT4-RAG-PHQ
Status: Enrolling by invitation | Type: Observational
Sponsor: University College, London (Other)
Responsible Party: Sponsor
Other Study IDs: 26133.001; 26133.001 (Other: UCL Research Ethics Committee)
Record Dates: First submitted 2025-01-24; First posted 2025-01-30 (Actual); Last update posted 2025-01-30 (Actual); Status verified 2025-01

CONDITIONS: Depression - Major Depressive Disorder; Depression Anxiety Disorder
Keywords: mental health; depression; chatbot; GPT; PHQ-9; RAG
MeSH Terms: conditions — Psychological Well-Being; Depression

STUDY DESIGN:
Observational Model: Other | Time Perspective: Cross-Sectional
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Procedure: GPT-4o and RAG Voice Chatbot for PHQ-9 Screening — This study involves the use of a voice-based chatbot powered by GPT-4o and Retrieval-Augmented Generation (RAG) to conduct depression screening using the Patient Health Questionnaire-9 (PHQ-9).
  The chatbot aims to evaluate the feasibility and acceptability of using AI-powered conversational tools for mental health screening.
  Participants interact with the chatbot in a single session, answering PHQ-9 questions and receiving responses generated using GPT-4o and RAG technologies.

SUMMARY:
This study aims to assess the feasibility and acceptability of a voice-based chatbot, powered by GPT-4o and Retrieval-Augmented Generation (RAG), for conducting depression screening using the Patient Health Questionnaire-9 (PHQ-9). The PHQ-9 is a validated self-report instrument widely used to screen, diagnose, and monitor the severity of depression. It consists of nine questions that correspond to the Diagnostic and Statistical Manual of Mental Disorders (DSM-5) criteria for major depressive disorder. Respondents rate the frequency of symptoms experienced over the past two weeks on a scale from 0 ("not at all") to 3 ("nearly every day"). The total score (ranging from 0 to 27) indicates the severity of depressive symptoms, categorized into minimal, mild, moderate, moderately severe, or severe depression. The PHQ-9 is also used to assess functional impairment and guide treatment decisions in clinical and research settings.

The voice-based chatbot integrates GPT-4o, with RAG to enhance its ability to provide informed and contextualized responses during interactions. GPT-4o serves as the conversational engine, capable of generating human-like, empathetic, and contextually appropriate dialogue. RAG, on the other hand, enables the chatbot to retrieve and incorporate external, up-to-date knowledge from a curated database or knowledge repository, ensuring the accuracy and reliability of its responses.

DETAILED DESCRIPTION:
Depression is a prevalent mental health challenge with significant personal, social, and economic costs. Traditional mental health resources face barriers such as stigma, limited availability, and long wait times. Technology, particularly AI-powered tools, provides an opportunity to bridge these gaps. This study utilizes GPT-4o and RAG to create a voice-interactive chatbot capable of conversational engagement, administering the PHQ-9 questionnaire, and delivering personalized feedback.

Participants will fill in the PHQ-9 for self-testing before interacting with the chatbot (the results will not be disclosed to the public and will only be used for accuracy comparisons), and the results of their self-tests will be compared with the results given by the chatbot in terms of accuracy.

The chatbot interaction comprises three phases:

1. Warm-up conversations for rapport-building and general support.

   * The chatbot initiates casual, empathetic dialogues to build rapport with users, helping them feel comfortable and at ease before transitioning to the PHQ-9 screening.
   * Users can ask general questions related to mental health, and the chatbot provides informed and supportive responses.
2. Administration of the PHQ-9 questionnaire for depression screening.

   * The chatbot introduces the PHQ-9 questionnaire, explaining its purpose and how the results will help assess the user's mental health.
   * Through voice interaction, users respond to the nine PHQ-9 questions, and the chatbot records their responses. The chatbot can clarify questions or provide additional context if users have difficulty understanding specific items.
3. Analysis of results and delivery of tailored recommendations.

   * After the user completes the PHQ-9, the chatbot analyzes the responses, calculates the total score, and categorizes the results into severity levels (e.g., mild, moderate).
   * Based on the score, the chatbot provides personalized recommendations, such as self-help strategies for mild symptoms or suggesting professional mental health services for more severe cases.

Participants will interact with the chatbot and then participate in a 1-hour semi-structured interview to provide feedback on their experience. The study focuses on evaluating the acceptability and feasibility of using such LLM-based chatbots in mental health screening and identifying potential improvements and risks.

Study Objectives Primary Objectives

1. To evaluate the acceptability, feasibility, and accuracy of a GPT-4o and RAG-based voice chatbot (HopeBot) for depression screening using PHQ-9.

   Hypothesis: Participants showed high acceptance of HopeBot (higher than 65%) and high willingness to use such LLM-based chatbot for mental health screening in the future (higher than 65%), indicating recognition of the credibility of LLM as a supportive tool in mental health screening (higher than 65%). Participants use of the HopeBot for depression screening matched their self-test PHQ-9 results by 100%
2. To analyze the chatbot's effectiveness in identifying depressive symptoms and delivering actionable recommendations.

Hypothesis: HopeBot can help users take the PHQ-9 test in a friendly way, help users categorize the answers accurately, and give accurate test results, the advice they provide is based on the official PHQ-9 guidelines, and more than 70% of the users say that their responses are very effective and helpful.

Secondary Objectives

1. To assess the feasibility and performance of integrating RAG with LLM in creating a voice-interactive chatbot for mental health.

   Hypothesis: Over 65% of participants recognized that responses using RAG were more helpful and effective.
2. To explore the strengths, limitations, and risks of deploying LLMs in the mental health domain.

Hypothesis: More than 65% of users say that HopeBot is very convenient, more accessible, and cost-free to provide non-judgmental advice. However, 50% still expressed concerns about its privacy and data security.

ELIGIBILITY:
Inclusion Criteria:

* Adults aged 18-65 years.
* Fluent in English.
* Access to a device capable of voice interaction and stable internet connection.
* Willing to participate in chatbot interaction and a follow-up interview.

Exclusion Criteria:

* Current severe psychiatric diagnoses (e.g., psychosis, bipolar disorder).
* Participants undergoing active treatment for depression with a psychiatrist.
* Discomfort with voice-based technology or inability to provide informed consent.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: The study population consists of healthy individuals aged 18 to 65 years who do not have severe mental illnesses. We welcome participants who have an interest in artificial intelligence technologies. Recruitment will be conducted both online and offline.
  Participants will engage with a sophisticated AI chatbot designed to simulate a consultation with a mental health professional. This interaction enables them to complete a psychometric evaluation, such as the PHQ-9 test, in a structured yet conversational manner. Unlike conventional online versions of the PHQ-9 test, the chatbot offers enhanced interactivity. For individuals who may experience difficulties in articulating or summarizing their responses, the chatbot provides clarifications and assistance using a comprehensive language model.
  After the assessment, participants will receive an interpretation of their test results along with tailored advice, delivered in accordance with established mental health guidelines.
Sampling Method: Non-Probability Sample
Enrollment: 100 (Estimated)
Dates: Start 2025-02-01 (Estimated); Primary Completion 2025-03-31 (Estimated); Study Completion 2025-05-31 (Estimated)

PRIMARY OUTCOMES:
Feasibility and Acceptability of the GPT-4o and RAG Voice Chatbot | Interviews are conducted immediately following the chatbot interaction.
  Participants' perceptions of the chatbot's feasibility, acceptability, and effectiveness are assessed through semi-structured interviews conducted after the interaction session. These interviews explore themes such as the chatbot's empathy, usability, and the overall user experience.

SECONDARY OUTCOMES:
Accuracy of PHQ-9 Scoring by the Chatbot | Measured immediately after the interaction session, once the chatbot has generated PHQ-9 scores
  The accuracy of the PHQ-9 scores generated by the chatbot is measured by comparing the chatbot's results to participants' self-reported PHQ-9 scores collected prior to the interaction. Agreement will be assessed using statistical methods such as Cohen's kappa or intraclass correlation coefficient (ICC).

CONTACTS AND LOCATIONS:
Overall Officials: Kezhi Li, Study Director — University College, London
Locations (1):
- UCL Institute of Health Informatics, London, United Kingdom

IPD SHARING:
Plan to Share IPD: No
IPD will not be shared to ensure participant confidentiality and comply with ethical guidelines related to mental health research. Additionally, participants did not provide explicit consent for data sharing with external researchers.